CLINICAL TRIAL: NCT04777903
Title: The Relationship Between Pre-pregnancy Body Mass Index (BMI) and Pregnancy Weight Gain and Pregnancy Outcomes in Women With Twin Pregnancy
Brief Title: The Relationship Between Pre-pregnancy BMI and Weight Gain and Outcomes in Women With Twin Pregnancy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: SAHoWMU-CR2021-07-201
Record Dates: First submitted 2021-02-28; First posted 2021-03-02 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Twin Pregnancy; Body Mass Index; Weight Gain; Pregnancy Outcome
MeSH Terms: conditions — Weight Gain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- underweight woman with twin pregnancy: underweight (BMI < 18.5 kg/m2)
  Interventions: Other: collect date about all participants
- normal weight woman with twin pregnancy: normal (BMI: 18.5-23.9 kg/m2)
  Interventions: Other: collect date about all participants
- overweight and obese woman with twin pregnancy: overweight and obese (BMI ≥24 kg/m2)
  Interventions: Other: collect date about all participants

INTERVENTIONS:
Other: collect date about all participants — a standardized and structured questionnaire that included information on age, residence, education, pregnancy history, disease history, height, and conception method, after obtaining the consent of all participants.

SUMMARY:
Prepregnancy body mass index (BMI) and gestational weight gain (GWG) have Significant effects on the risk of pregnancy outcomes such as gestational hypertension disease and gestational diabetes mellitus in singleton pregnancies. This paper is to investigate the relationship between pre-pregnancy body mass index (BMI) and weight gain during pregnancy and pregnancy outcomes in women with twin pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 ~ 41 years old;
* The gestational age of the first diagnosed twin pregnancy is ≤10weeks;
* Double chorionic double amniotic sac pregnancy;

Exclusion Criteria:

* with heart disease, liver disease, kidney disease, complications (chronic hypertension, hyperthyroidism, diabetes and others ), genetic diseases, psychological and mental diseases;
* with history of habitual abortion and cervical insufficiency;

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Eligible participants is female.
Study Population: The participants include women with twin pregnancy meeting the inclusion criteria
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
the incidence of gestational diabetes mellitus, gestational hypertension and small for gestational age | 35 weeks to 40 weeks gestation
  pregnant outcome

CONTACTS AND LOCATIONS:
Overall Officials: Ying Hua, Study Director — Second Affiliated Hospital of Wenzhou Medical University
Locations (1):
- department of obstetrics of Second Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China